CLINICAL TRIAL: NCT05852769
Title: A Phase 1, Single-center, Open-label, Sequential Study to Evaluate the Drug-drug Interaction Potential of BMS-986196 in Healthy Participants
Brief Title: A Study to Evaluate the Drug-drug Interaction Potential of BMS-986196 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IM038-022
Record Dates: First submitted 2023-05-01; First posted 2023-05-10 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Healthy Volunteers
Keywords: BMS-986196
MeSH Terms: interventions — Caffeine; montelukast; Flurbiprofen; Omeprazole; Midazolam; Digoxin; Pravastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BMS-986196 and/or Cocktail Probe Substrate Drugs (Experimental)
  Interventions: Drug: BMS-986196; Drug: Caffeine; Drug: Montelukast; Drug: Flurbiprofen; Drug: Omeprazole; Drug: Midazolam; Drug: Digoxin; Drug: Pravastatin

INTERVENTIONS:
Drug: BMS-986196 — Specified dose on specified days
Drug: Caffeine — Specified dose on specified days
Drug: Montelukast — Specified dose on specified days
Drug: Flurbiprofen — Specified dose on specified days
Drug: Omeprazole — Specified dose on specified days
Drug: Midazolam — Specified dose on specified days
Drug: Digoxin — Specified dose on specified days
Drug: Pravastatin — Specified dose on specified days

SUMMARY:
This study is designed to assess the effect of BMS-986196 on the drug levels of caffeine, montelukast, flurbiprofen, omeprazole, midazolam, digoxin, and pravastatin in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations.
* Body mass index of 18.0 to 33.0 kilogram per meter squared (kg/m^2), inclusive, and body weight ≥50.0 kg.

Exclusion Criteria:

* History of rhabdomyolysis.
* History of peptic ulcer disease or significant GI bleeding.
* History of malignancy in the 5 years prior to screening (except fully excised basal cell carcinoma).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 26 days
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC[INF]) | Up to 26 days
Area under the plasma concentration-time curve from time zero to time of the last quantifiable concentration (AUC[0-T]) | Up to 26 days

SECONDARY OUTCOMES:
Time of maximum observed serum concentration (Tmax) | Up to 26 days
Apparent terminal phase half-life (T-Half) | Up to 26 days
Apparent total body clearance (CLT/F) | Up to 26 days
Number of participants with adverse events (AEs) | Up to 52 days
Number of participants with vital sign abnormalities | Up to 28 days
Number of participants with electrocardiogram (ECG) abnormalities | Up to 21 days
Number of participants with physical examination abnormalities | Up to 28 days
Number of participants with clinical laboratory abnormalities | Up to 28 days
Intensity of Suicidal Ideation as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) Score | Up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- ICON plc, Millcreek, Utah, United States

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com